CLINICAL TRIAL: NCT01531166
Title: An Observational, Multi-Center, Cohort Study Evaluating the Antiviral Efficacy, Safety, and Tolerability in Korean Patients With Chronic Hepatitis B (CHB) Receiving Pegylated Interferon-alpha 2a (Pegasys®): TRACES STUDY
Brief Title: A Cohort Study in Korean Patients With Chronic Hepatitis B (CHB) Receiving Pegylated Interferon
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2011-0461
Record Dates: First submitted 2012-01-31; First posted 2012-02-10 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Chronic Hepatitis B
Keywords: Chronic hepatitis B; pegylated Interferon-alpha 2a; Korean
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon alfa-2a

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Chronic hepatitis B
  Interventions: Drug: pegylated Interferon-alpha 2a

INTERVENTIONS:
Drug: pegylated Interferon-alpha 2a — Pegasys 180mcg/PFS/ subcutaneous injection / Once a week
  Other Names: Pegasys

SUMMARY:
The current proposed study aims to bring answers following issues: the antiviral efficacy and safety profiles in Korean Chronic Hepatitis B (CHB) patients who are mostly infected with solely genotype C HBV, a proper duration of Pegasys® therapy post-treatment durability or accumulation of HBeAg seroconversion/HBsAg loss, preventable effect on long-term disease progression to liver cirrhosis and liver cancer. In addition, this study aims to collect more data on the efficacy and safety in a real-life clinical setting of Pegasys® therapy in patients with CHB.

DETAILED DESCRIPTION:
* Korea is known to be an endemic area for HBV infection. Some studies have reported that more than 95% of patients in Korea with chronic HBV have genotype C infection.
* Compared with other genotypes, genotype C is associated with increased viral loads, higher histologic activity, more severe acute exacerbations, a longer viral clearance phase and worse antiviral response to peg-interferon therapy.
* Long-term nucleos(t)ide analogue (NA) therapy is recommended for chronic hepatitis B (CHB) patients with compensated and decompensated liver disease. However, a possibility of cessation of antiviral treatment with oral NAs is unlikely due to rebound of HBV DNA levels after termination of NAs administration. In addition, NA therapy has been reported to have lower chance of HBsAg seroclearance compared to that with immunomodulatory agents such as peginterferon.
* Pegasys® has been proved to induce HBsAg loss, which is the closest to cure of disease. However, a better understanding of HBV treatment with Pegasys® in the real-life clinical setting in Korea can be helpful for decision of treatment strategy in the future. Asian experience with Pegasys® therapy in CHB is limited. Study populations of investigator-initiated trials consist of selected group with smaller number of Korean patients. Therefore, long-term efficacy and safety data in real practice with Pegasys® treatment in both HBeAg-positive and -negative Korean patients are necessary.
* In addition, the current proposed collected data study may be helpful to bring answers to many unresolved issues: the antiviral efficacy and safety profiles in Korean CHB patients who are mostly infected with solely genotype C HBV, a proper duration of Pegasys® therapy post-treatment durability or accumulation of HBeAg seroconversion/HBsAg loss, preventable effect on long-term disease progression to liver cirrhosis and liver cancer. In addition, this study aims to collect more data on the efficacy and safety in a real-life clinical setting of Pegasys® therapy in patients with CHB.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects receiving treatment for CHB with PEGASYS according to standard of care and in line with the current summary of product characteristics(SPC)/ local labeling who have no contra-indication to PEGASYS therapy as per the local label.
* Adult chronic hepatitis B patients (20 years of age or older) who has been completed or are currently receiving or are planned to receive Pegasys® as a first-line therapy.
* Those with baseline HBV DNA > 2,000 IU/mL and elevation of ALT level.
* HBeAg positive or HBeAg negative serologically proven chronic hepatitis B(CHB)
* Subjects treated with previous NAs therapy are eligible for this study.

Exclusion Criteria:

Subjects with ALT > 10 x ULN or evidence of hepatocellular carcinoma.

* Subjects should be without serological evidence of co-infection with HCV, HIV, or HDV.
* Subjects with decompensated liver disease, as well as pregnant or breast-feeding women, will not be eligible for the study.
* Subjects should have no other diseases that might be contraindication to peg-interferon therapy as per local SPC (e.g., severe psychiatric diseases, immunological diseases, severe retinopathy or thyroid dysfunction, history of severe pre-existing cardiac disease, etc)
* Subjects with other contra-indications to PEGASYS therapy as detailed in the label (hypersensitivity to the active substance, to alpha interferons, or to any of the excipients)
* A history of liver transplantation or planned for liver transplantation
* Subjects who receive concomitant therapy with telbivudine.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HBeAg-positive and HBeAg-negative chronic hepatitis B patients who have completed or are currently on Pegasys® monotherapy as a first line therapy. In addition, all consecutive CHB patients who will be initiated on Pegasys® in 2011 will be prospectively enrolled.
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2011-09; Primary Completion 2014-08 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
HBsAg loss or appearance of anti-HBs antibody in treatment-naïve Korean CHB patients treated with Pegasys | 2015 (up to 3 years)

SECONDARY OUTCOMES:
Sustained suppression of HBV DNA | 2015 (up to 3 years)
HBeAg loss and seroconversion in HBeAg-positive CHB | 2015 (up to 3 years)
ALT normalization | 2015 (up to 3 years)

CONTACTS AND LOCATIONS:
Overall Officials: Sang Hoon Ahn, MD. PhD, Study Chair — Department of Internal Medicine, Yonsei Universtiy College of Medicine,
Locations (1):
- Sang Hoon Ahn, Seoul, Seodaemun-gu, South Korea